CLINICAL TRIAL: NCT05085249
Title: Improving Goal Directed Medical Therapy for Device Clinic Patients With Reduced Ejection Fraction at the University of Ottawa Heart Institute: a Quality Improvement Initiative (VIGILANT)
Brief Title: Improving Goal Directed Medical Therapy for Device Clinic Patients With Reduced EF at UOHI: a QI Initiative (VIGILANT)
Acronym: VIGILANT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Novartis (Industry); Servier (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mehrdad Golian, Cardiologist, Ottawa Heart Institute Research Corporation
Other Study IDs: 2021_Vigilant_QA
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: Quality assurance; Medication optimization; Device clinic; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a quality improvement initiative with the goal of optimizing heart failure (HF) patients seen through the outpatient cardiac implantable electronic device clinic at the University of Ottawa Heart Institute (UOHI). The UOHI device clinic oversees more than 12,000 in-clinic patient visits annually with over 5000 visits for patients with reduced ejection fraction (EF) and HF. In patients with reduced EF, guideline directed medical therapy compliance (GDMT) is sub-optimal in real world clinical practice. Considering the most recent changes to The Canadian Cardiovascular Society heart failure guideline recommendations, the compliance rate may be even lower than reported rates in the literature.

The goal of this study is to optimize GDMT through collaboration between the HF clinic, a HF/arrhythmia nurse practitioner, and application of a nurse run algorithm based pathway to identify patients suitable for medication optimization and guiding the most responsible physician (MRP) for their heart failure (PCP, cardiologist or HF physician) through a letter. The compliance rate will also be re-evaluated to assess improvement in GDMT in this patient population. GDMT will ensure the greatest chance to improve patient outcomes by reducing heart failure hospitalizations, emergency room visits, ventricular arrhythmias, implantable cardioverter defibrillator shocks, clinic visits, and thereby improving patients' quality of life.

DETAILED DESCRIPTION:
The goal of this quality improvement initiative is to optimize goal directed medical therapy compliance (GDMT) in heart failure (HF) patients seen at the University of Ottawa Heart Institute (UOHI) device clinic. GDMT is reported as low as 45% and a recent Canadian survey reports estimated compliance as low as 15%. The project will be performed in 3 phases. Phase 1 will aim to establish the rates of GDMT compliance in heart failure patients seen through the device clinic. The chart of 600 consecutive implantable cardioverter defibrillator (ICD) patients will be reviewed to establish the current compliance rate with GDMT in patients with reduced ejection fraction (EF). In Phase 2, the goal is to optimize GDMT through collaboration between the HF clinic and a nurse run algorithm based pathway to identify patients suitable for medication optimization and guiding the most responsible physician (MRP) for their heart failure (PCP, cardiologist or HF physician) through a letter. The ultimate goal is to improve the quality of life of patients seen at the institute. In Phase 3, the compliance rate will be re-evaluated every 6 months to assess for improvement in GDMT in this patient population.

During Phase 1 (establishing baseline medication compliance), the charts of 600 consecutive ICD patients will be reviewed using PACeART and EPIC databases. Rate of GDMT compliance will be calculated. For the purposes of this investigation, and in patients with EF < 40% at the time of ICD clinic visit, GDMT is defined as:

1. NHYA I and ACE-I/ARB OR ARNI+BB+MRA+SGL2 or
2. NYHA II or above and on ARNI+BB+MRA+SGL2

ACE-I refers to Angiotensin-converting-enzyme inhibitor medication, ARB refers to Angiotensin II receptor blocker medication, ARNI refers to angiotensin receptor neprilysin inhibitor medication, BB refers to beta blocker medication, MRA refers to aldosterone receptor antagonist medication, and SGL2 refers to sodium-glucose cotransporter-2 inhibitor medication.

During Phase 2 (medication optimization through collaborative work with heart function clinic, primary cardiologist and device clinic), all patients seen with ICD and reduced EF at the UOHI device clinic will be given a questionnaire by the clinic assistant. The questionnaire will be comprised of 2 questions:

1. Does ordinary physical activity (i.e. walking to the device clinic, grocery shopping, etc.) cause palpitation, fatigue, shortness of breath or chest pain? (yes/no)
2. Have you been admitted to the hospital for heart failure in the past year? (yes/no)

If patient has answered no to both questions of the survey they will be classified as NYHA I, all others will be classified as NYHA II or greater. Medication lists will be updated for all patients by the device clinic nurse in EPIC. Blood pressure and pulse will also be documented in EPIC by the device clinic nurse for all in-person appointments. A clinical nurse or physician assistant will review all patient visits for ICD and reduced EF at the UOHI device clinic, patients not on GDMT (defined above) will have a letter sent to their cardiologist with recommendations on medication change and required follow up. Those without a cardiologist will be referred to the heart function clinic at UOHI or general hospital for medication optimization. Patients will be categorized into 4 groups:

1. Patients on GDMT and at target dose (no action required)

   Those on GDMT will continue on the same medication with no change. In patients with EF < 40% at the time of ICD clinic visit, GDMT is defined as:
   1. NHYA I and ACE-I/ARB OR ARNI+BB+MRA+SGL2 or
   2. NYHA II or above and on ARNI+BB+MRA+SGL2
2. Patients that require up titration of medication. These patients have been identified as NYHA II or above and they are not on the target dose of medication. A quality officer reviews the answers to the questionnaire, their current medications, and if systolic blood pressure > 100 mmHg. a letter of will be sent to the pts cardiologist and a copy will be given to the patient regarding medication optimization recommendation and required follow up. Medication doses and required follow up will be detailed in the letter.
3. Patient requires a change in medication but has not cardiologist. A referral will be made by the nurse or physician's assistant to the UOHI heart function clinic for medication optimization for patients identified as NYHA II or above and require initiation of ANRI, SGL2, BB, or MRA. Blood requisition will also be given to and results will be sent to the referred MD. All patients who have their medication increased or referred to have their medication switched and up titrated through the heart function medication optimization clinic will have a letter sent to their care team (cardiologist and family physician) informing them of the referral and change in medication.
4. Patients already actively followed by the HF clinic will have an appointment made with their HF cardiologist.

During Phase 3 (re-evaluation), patients will bring the letter from their cardiologist stating the reason why they were not started on the recommended medication (i.e. renal function, patient preference, urinary tract infection, low blood pressure, hyperkalemia etc.). The medication use will be rated every 6 months through EPIC to assess for increase in medication uptake. In addition, annually 35 (approximately 10% of the ICD implants) randomly selected ICD patients with reduced ejection fraction from the device clinic will be assessed regarding GDMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with implantable cardioverter-defibrillator
* Ejection fraction ≤ 35%

Exclusion Criteria:

* None (QA project)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen at the University of Ottawa Heart Institute electronic device clinic who have an implantable cardioverter defibrillator device. Patients served are primarily from Ottawa and the surrounding region. As a tertiary care centre, UOHI also sees referrals from other regions across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Goal directed medical therapy compliance | 6 months
  Rate of compliance will be assessed in this initiative

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Golian, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No